CLINICAL TRIAL: NCT02350192
Title: A Randomized Controlled Trial of the Effectiveness of a Home-based Interactive E-health Educational Intervention for Middle-aged Cardiovascular Disease Adults in Improving Total Exercise, Adherence Rate, Exercise Efficacy and Outcomes
Brief Title: Effectiveness of an E-health Educational Intervention for Cardiovascular Disease Adults in Improving Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Mi Ling Eliza, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10110301
Record Dates: First submitted 2015-01-21; First posted 2015-01-29 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Disease
Keywords: ehealth; intervention; effectiveness; randomized controlled trial
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-health educational intervention (eHEI) (Experimental): Participants in the intervention group received usual care and additional individualized educational intervention administered by a trained nurse who was experienced in cardiac nursing. The exercise prescription had been set as walking exercise for 30 minutes per day for 5 days per week. The exercise dosage might be modified with physician's order to suit the individual's physical condition and agreed goals if necessary. The 30- minutes educational intervention was conducted in a private room of the clinic. The content covered general information related to coronary heart disease and benefit of performing exercise, the e-health educational intervention (eHEI) link demonstration and re-demonstration. In addition, one telephone follow-up was conducted at week 2 to facilitate the usage of the e-HEI link.
  Interventions: Behavioral: e-health educational intervention (eHEI)
- Control group (No Intervention): Control group received standard care only. The control group also received standard usual care comprising the doctor follow up with medication. During an individualized educational session conducted by a trained research assistant , a briefing on healthy life style and an an additional educational leaflet about coronary heart disease which is customarily given to patient with cardiovascular risks was given to the patient. In the control group, no e-health educational intervention has been provided to the patients of the control group.

INTERVENTIONS:
Behavioral: e-health educational intervention (eHEI) — The e-HEI link (e-health link http://ehealth.nur.cuhk.edu.hk) provides the content of culture-specific cognitive knowledge related to CVD and measures to modify risk factors. The member area and interactive platform of the e-HEI website allows the self-monitoring of individual health and exercise records. Members can view and retrieve their own exercise records daily, and health measures trend regularly.
  Arms: e-health educational intervention (eHEI)

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death globally and e-health educational programs have been proved to be effective support to CVD clients. However, most e-health programs lack personalization and this seldom results in exercise behavioral change. Considering the advantages of e-health programs, as well as the widespread internet use and the rising trend of younger patients having CVD in Hong Kong, we conducted a Randomized Controlled Trial (RCT) to investigate the effectiveness of a home-based interactive e-health educational intervention versus usual care for middle aged cardiac vascular (CV) patients on their total physical exercise, exercise adherence and quality of life.

DETAILED DESCRIPTION:
Introduction:

Cardiovascular disease (CVD) is the leading cause of death globally and e-health educational programs have been proved to be effective support to CVD clients. However, most e-health programs lack personalization and this seldom results in exercise behavioral change. Considering the advantages of e-health programs, as well as the widespread internet use and the rising trend of younger patients having CVD in Hong Kong, we conducted a Randomized Controlled Trial (RCT) to investigate the effectiveness of a home-based interactive e-health educational intervention versus usual care on total physical exercise, exercise adherence and self efficacy, risk factor profile, psychological outcomes and quality of life for middle aged cardiac vascular (CV) patients.

Methods and analysis:

This is a prospective randomised clinical trial investigating effectiveness of a home-based interactive e-health educational intervention for middle-aged cardiovascular disease (CVD) adults in improving total exercise, adherence rate, exercise efficacy and outcomes. The hypothesis is that the middle-aged CVD patients (those who are 40-65 years old) would be more likely to adhere to exercise-based behavior that improves their total exercise, exercise adherence rate, cardiac risk profile , psychological outcomes and quality of life with the support of an interactive e-health educational intervention.

The RCT was conducted in two government cardiac clinics in Hong Kong. 438 eligible CV clients were randomized to either the control group (C) or the intervention group (I) using block randomization method. All participants received usual care while (I) additionally received the e-health educational intervention (eHEI) programme. This programme comprised of one-hour educational session, one telephone follow up and e-health link on self monitoring including record of health measures and physical exercise across 6 months. Data was collected at baseline, three months and six months intervals. The primary outcome was total physical exercise (GSLTPAQ). Secondary outcomes consisted of: exercise efficacy and adherence rate; CV risk profile; physical and psychological health outcomes (SF12 & HAD); biological parameter. Data was analyzed using generalized linear models.

Ethics and dissemination: The study complies with the Declaration of Helsinki and was approved by the University and hospital ethics committee. Study findings will be disseminated in international conferences and publications.

Key messages:

Cardiovascular disease (CVD) is the leading cause of death globally and most e-health educational programs have been proved to be effective support to CVD clients. However, most e-health programs lack personalization and this seldom results in exercise behavioral change.

The adopted e-health program aims to empower CVD participants by increase knowledge on cardiovascular risks, perceived benefits of exercise to health, as well as enhance their self-efficacy in exercise adherence and exercise behavior. Data analysis has been started in August 2015. This trial will provide evidence of e-health programs on physical and psychological outcomes comprehensively.

Strengths and limitations of this study:

The study has been designed to meet the criteria for high quality in non-pharmacological randomised clinical trials with randomisation, multicentre participation, blinded assessment and analysis with good sample size.

ELIGIBILITY:
Inclusion Criteria:

* being an ethnic Chinese adult
* who attends regular follow-up treatments for their CVD problems
* aged 30-65
* able to use and access the internet at home
* willing to participate (with corresponding signed consent form)

Exclusion Criteria:

* those with physical, mental, visual, or cognitive impairments as recorded in their health records
* those who have contra-indications to walking.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in total physical exercise (measured by The Godin-Shephard Leisure-Time Physical Activity Questionnaire) | Baseline, 3 Months, 6 Months
  Change in physical exercise is

SECONDARY OUTCOMES:
Changes in exercise efficacy (measured by a validated scale. The scale consists of 9 items and responses are made on a 0-10 scale) | Baseline, 3 Months, 6 Months
  Changes in self-efficacy for exercise is measured by a validated scale. The scale consists of 9 items and responses are made on a 0-10 scale.
Exercise adherence (two simple questions will be asked: how often do you do any physical activity per week? and What is the duration of the exercise on average?) | Baseline, 3 Months, 6 Months
  To measure exercise adherence, two simple questions will be asked: how often do you do any physical activity per week? and What is the duration of the exercise on average?
Changes in anxiety and depression (Chinese version of the Hospital anxiety and depression scale) | Baseline, 3 Months, 6 Months
  The Chinese version of the Hospital anxiety and depression scale will be used to measure the changes in anxiety and depression. The scale consists of 14 items and responses on a 4 point likert scale.
Changes in quality of Life (Chinese version of the health survey questionnaire (SF-12) | Baseline, 3 Months, 6 Months
  Chinese version of the health survey questionnaire (SF-12) will be used in measuring the changes in quality of life.
Cardiac risk factor profile (Demographic data will be collected through questionnaire) | Baseline, 3 Months, 6 Months
  Demographic data will be collected through questionnaire. Medical problems, cardiac risk profile such as (systolic and diastolic blood pressure, LDL cholesterol, HDL cholesterol, triglycerides, blood sugar level, HbA1c, BMI will be retrieved from the patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Mi Ling Wong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Tung Wah Eastern Hospital, Causeway Bay, Hong Kong Island
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong Island

IPD SHARING:
Plan to Share IPD: No